CLINICAL TRIAL: NCT02580110
Title: On the Impact of Common Sweetening Agents on Glucose Regulation, Cognitive Functioning and Gut Microbiota
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: Anti-Diabetic Food Centre (Other)
Responsible Party: Principal Investigator, Anne Nilsson, PhD, assocoate professor, Lund University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 2015/57
Record Dates: First submitted 2015-10-14; First posted 2015-10-20 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-06

CONDITIONS: Healthy Subjects
Keywords: no specific condition
MeSH Terms: interventions — Sucrose; Saccharin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- sucrose (Experimental): 14 days intervention with daily intake of a beverage (1000 ml) including 66g sucrose.
  Interventions: Other: Sucrose
- stevia glycosides (Experimental): 14 days intervention with daily intake of a beverage (1000ml) including 0.220 g stevia glycosides.
  Interventions: Other: Stevia glycosides
- saccharin (Experimental): 14 days intervention with daily intake of a beverage (1000ml) including 0.216g saccharin.
  Interventions: Other: saccharin

INTERVENTIONS:
Other: Sucrose
  Arms: sucrose
Other: Stevia glycosides
  Arms: stevia glycosides
Other: saccharin
  Arms: saccharin

SUMMARY:
The study intention is to investigate, in healthy humans, effects of 3 commonly used sweeteners on cardiometabolic risk markers, cognitive functions, and influences on gut microbiota composition.

DETAILED DESCRIPTION:
Healthy subjects will be included in a crossover study with the purpose to investigate effects of 3 commonly used sweeteners on cardiometabolic risk markers, cognitive functions, and influences on gut microbiota composition. The subjects will consume each test product for 14 days in a random order, separated by at least a two-week washout period. On the last day in each intervention period, i.e. at day fifteen, the last test portion will be consumed together with a standardized evening meal at 9.00 pm. Thereafter the subjects are fasting until arriving to the experimental unit. Upon arrival, test variables in blood will be determined at fasting and repeatedly for 3h postprandial a standardised breakfast served approximately at 8.00 am. Cognitive performance will be determined in the postprandial period with tests evaluating working memory capacity, selective attention, psychomotor reaction time, and executive functions. After each intervention period, faecal samples will be collected for characterization of gut microflora.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects
* blood glucose <6.1
* BMI <28
* age between 40-70 years
* normal diet
* fluent in Swedish language (due to the structure of the cognitive tests).

Exclusion Criteria:

* diabetes
* cognitive decline (not able to cope with the cognitive tests)
* metabolic syndrome
* gastro-intestinal disorders
* antibiotics or probiotics during the study period
* smookers

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2015-10; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Incremental area under the curve (iAUC) (Glucose tolerance) | predose (standardised breakfast), 0, 15, 30, 45, 60, 90, 120, 150, and 180 min post dose.
  The iAUC are determined after a standardized breakfast based on white wheat bread (50g available starch). The breakfast was commenced at time=0 and consumed within 10-12 min.
Incremental area under the curve (iAUC) (insulin sensitivity). | predose, 0 (fasting), 15, 30, 45, 60, 90, 120, 150, and 180 min post-dose.
  The iAUC are determined after a standardized breakfast based on white wheat bread (50g available starch). The breakfast was commenced at time=0 and consumed within 10-12 min.
Working memory capacity | 80 min after the standardised breakfast
  Working memory capacity determined with an oral working memory test composed of short sentences that can be semantically meaningful or not. 3-5 sentences are read to the subject. After each sentence the subject immediately has to reply if the sentence is semantically meaningful or not. After the set of 3-5 sentences the subjects have to recall the first noun in each of the sentences. One test is composed of 12 set with (3-5) sentences.
Glut microbiota composition | baseline and after 14 days intervention
  faecal samples are collected at baseline prior to the study and after each 14 day intervention period
Working memory capacity | 120 min
  Working memory capacity determined with an oral working memory test composed of short sentences that can be semantically meaningful or not. 3-5 sentences are read to the subject. After each sentence the subject immediately has to reply if the sentence is semantically meaningful or not. After the set of 3-5 sentences the subjects have to recall the first noun in each of the sentences. One test is composed of 12 set with (3-5) sentences.
Working memory capacity | 160 min
  Working memory capacity determined with an oral working memory test composed of short sentences that can be semantically meaningful or not. 3-5 sentences are read to the subject. After each sentence the subject immediately has to reply if the sentence is semantically meaningful or not. After the set of 3-5 sentences the subjects have to recall the first noun in each of the sentences. One test is composed of 12 set with (3-5) sentences.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Nilsson, PhD, Principal Investigator — Food for Health Science Centre, Lund University
Locations (1):
- Food for Health Science Centre, Medicon Village, Lund University, Lund, Sweden